CLINICAL TRIAL: NCT04660331
Title: PROMOTE Pilot Study: Pharmacy Multimodal Communication Strategy to Promote HPV Vaccination
Brief Title: Communication Strategy to PROMOTE HPV Vaccination in Pharmacies: PROMOTE Study
Acronym: PROMOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Parth Shah, Assistant Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1007825; NCI-2020-08529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10600 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-12-09 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Delivery of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim I (interview) (Experimental): Participants participate in a semi-structured interview in-person or via phone over 90 minutes about barriers/facilitators of HPV vaccination in pharmacies.
  Interventions: Behavioral: Healthcare Activity
- Aim 2 (survey, training, communication intervention, and environmental scan) (Experimental): Participants provide feedback on survey questions via cognitive testing. Pharmacy staff complete an online survey over 10-15 minutes to assess the acceptability, appropriateness, and feasibility of providing HPV vaccination to children aged 9-17 in their pharmacies. Pharmacy staff then attend two, 60- minute vaccine communication training sessions, consisting of identifying vaccine-eligible children and recommending HPV and other vaccines. Pharmacy staff employ the new communication strategy in their pharmacy up to 6 months, and then complete an online survey over 10-15 minutes.
  Pharmacies of which the pharmacy staff participants work undergo an environmental scan to characterize the pharmacy's environment, vaccination workflow, and team dynamics.
  Interventions: Other: Communication Intervention; Other: Communication Skills Training; Behavioral: Healthcare Activity; Other: Survey Administration

INTERVENTIONS:
Other: Communication Intervention — Undergo communication strategy intervention
  Arms: Aim 2 (survey, training, communication intervention, and environmental scan)
Other: Communication Skills Training — Undergo communication training sessions
  Arms: Aim 2 (survey, training, communication intervention, and environmental scan)
Behavioral: Healthcare Activity — Participate in interview
  Other Names: Health Care Activity; Healthcare
  Arms: Aim I (interview)
Behavioral: Healthcare Activity — Undergo environmental scan
  Other Names: Health Care Activity; Healthcare
  Arms: Aim 2 (survey, training, communication intervention, and environmental scan)
Other: Survey Administration — Complete survey
  Arms: Aim 2 (survey, training, communication intervention, and environmental scan)

SUMMARY:
This trial investigates how a communication strategy works in increasing human papillomavirus (HPV) vaccines in community pharmacies among adolescents. Although pharmacies are vaccine providers, low vaccination rates are persistent as a result of low awareness of pharmacy services and poor engagement by pharmacy staff with adolescents about vaccines. The purpose of this study is to test a communication strategy that identifies vaccine-eligible children and teaches pharmacy staff how to effectively communicate with them about HPV vaccination in order to increase HPV vaccination rates.

DETAILED DESCRIPTION:
OUTLINE:

AIM 1: Participants participate in a semi-structured interview in-person or via phone over 90 minutes about barriers/facilitators of HPV vaccination in pharmacies.

AIM 2: Participants provide feedback on survey questions via cognitive testing. Pharmacy staff complete an online survey over 10-15 minutes to assess the acceptability, appropriateness, and feasibility of providing HPV vaccination to children aged 9-17 in their pharmacies. Pharmacy staff then attend two, 60-minute vaccine communication training sessions, consisting of identifying vaccine-eligible children and recommending HPV and other vaccines. Pharmacy staff employ the new communication strategy in their pharmacy up to 6 months, and then complete an online survey over 10-15 minutes.

Pharmacies of which the pharmacy staff participants work undergo an environmental scan to characterize the pharmacy's environment, vaccination workflow, and team dynamics.

Additionally, pharmacy audits will be conducted from the pharmacy electronic records to assess adoption of HPV vaccination, and the impact of the communication strategy on adoption of other adolescent vaccines (e.g., tetanus, diphtheria, acellular pertussis; meningococcal conjugate; influenza).

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 (PARENTS/GUARDIANS): Individuals with children between the ages of 9-17 in their care who are English speakers, live in Washington state, and have access to a telephone or computer with internet access (up to 12 parents)
* AIM 1 (PHARMACY STAFF): Employed at a Western Washington Bartell Drugs pharmacy sites and have access to a telephone or computer with internet access
* AIM 2: Pharmacy staff employed at up to four independent pharmacies in western Washington state who speak English and have access to a computer with internet access

Exclusion Criteria:

* AIM 1 (PARENTS/GUARDIANS): Those who object to having their interview audio recorded
* AIM 1 and AIM 2 (PHARMACY STAFF): Floaters/per diem. Those who object to having their interview audio recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PROMOTE Key Informant Interviews: Parents/Guardians (Aim 1): Participants in the key informant interview phase (Aim 1) whose goal was to adapt an existing electronic forecasting system and behavioral counseling framework to match barriers and facilitators to HPV vaccination in pharmacies, administered by the Principal Investigator. Participants are parents/guardians of children aged 9-17 in Western Washington.
  Key informant interviews were conducted with the participants described above using semi-structured interview techniques and guided by theoretical domain framework.
  Interviews were conducted by trained study staff members over the phone and lasted approximately 90 minutes. The interview included demographic survey questions.
- PROMOTE Key Informant Interviews: Pharmacy Staff (Aim 1): Participants in the key informant interview phase (Aim 1) whose goal was to adapt an existing electronic forecasting system and behavioral counseling framework to match barriers and facilitators to HPV vaccination in pharmacies, administered by the Principal Investigator. Participants are pharmacy staff in Western Washington.
  Key informant interviews were conducted with the participants described above using semi-structured interview techniques and guided by theoretical domain framework.
  Interviews were conducted by trained study staff members over the phone and lasted approximately 90 minutes. The interview included demographic survey questions.
- PROMOTE Intervention (Aim 2): Participants in the intervention group an adapted multi-modal communication strategy to support HPV vaccination in pharmacies administered by the Principal Investigator. Participants are pharmacy staff in Western Washington.
  The intervention consists of a multi-modal strategy that includes adapting an existing electronic "forecasting" system to identify vaccine eligible children who are due for vaccination and communication training for pharmacy staff to effectively recommend HPV vaccination.
  The intervention was delivered in one 60-minute session recorded and available online as a continuing education training that covered five modules: 1) educational overview of adolescent vaccination, 2) overview of the communication strategy, 3) process for integrating the strategy into clinical workflow, 4) training on communication strategy, and 5) pharmacy staff practice of the strategy.
Period: PROMOTE Key Informant Interviews (Aim 1)
Arm/Group | PROMOTE Key Informant Interviews: Parents/Guardians (Aim 1) | PROMOTE Key Informant Interviews: Pharmacy Staff (Aim 1) | PROMOTE Intervention (Aim 2)
Started | 13 | 11 | 0
Completed | 13 | 11 | 0
Not Completed | 0 | 0 | 0
Period: PROMOTE Intervention (Aim 2)
Arm/Group | PROMOTE Key Informant Interviews: Parents/Guardians (Aim 1) | PROMOTE Key Informant Interviews: Pharmacy Staff (Aim 1) | PROMOTE Intervention (Aim 2)
Started | 0 | 0 | 18
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Participants in the two Aim 1 arms are English-speaking pharmacy staff and parents or guardians of children aged 9-17. Participants in the Aim 2 arm are English-speaking pharmacy staff at enrolled sites participating in a remote, 1-part communication strategy intervention. There is no participant overlap between the groups.
Groups:
- PROMOTE Aim 1 Interviews: Pharmacy Staff: Participants in the key informant interview phase (Aim 1) whose goal was to adapt an existing electronic forecasting system and behavioral counseling framework to match barriers and facilitators to HPV vaccination in pharmacies, administered by the Principal Investigator. Participants are pharmacy staff and in Western Washington.
  Key informant interviews were conducted with the participants described above using semi-structured interview techniques and guided by theoretical domain framework.
  Interviews were conducted by trained study staff members over the phone and lasted approximately 90 minutes. The interview included demographic survey questions.
- PROMOTE Aim 1 Interviews: Parents: Participants in the key informant interview phase (Aim 1) whose goal was to adapt an existing electronic forecasting system and behavioral counseling framework to match barriers and facilitators to HPV vaccination in pharmacies, administered by the Principal Investigator. Participants are parents/guardians of children aged 9-17 in Western Washington.
  Key informant interviews were conducted with the participants described above using semi-structured interview techniques and guided by theoretical domain framework.
  Interviews were conducted by trained study staff members over the phone and lasted approximately 90 minutes. The interview included demographic survey questions.
- PROMOTE Aim 2 Intervention: Participants in the intervention group an adapted multi-modal communication strategy to support HPV vaccination in pharmacies administered by the Principal Investigator. Participants are pharmacy staff in Western Washington.
  The intervention consists of a multi-modal strategy that includes adapting an existing electronic "forecasting" system to identify vaccine eligible children who are due for vaccination and communication training for pharmacy staff to effectively recommend HPV vaccination.
  The intervention was delivered in one 60-minute session recorded and available online as a continuing education training that covered five modules: 1) educational overview of adolescent vaccination, 2) overview of the communication strategy, 3) process for integrating the strategy into clinical workflow, 4) training on communication strategy, and 5) pharmacy staff practice of the strategy.
- Total: Total of all reporting groups
Arm/Group | PROMOTE Aim 1 Interviews: Pharmacy Staff | PROMOTE Aim 1 Interviews: Parents | PROMOTE Aim 2 Intervention | Total
Number analyzed (Participants) | 11 | 13 | 18 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8.6) | 44.5 (5.1) | 44.17 (13.01) | 39.89 (7.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex, Female | 6 | 13 | 11 | 30
  Sex, Male | 5 | 0 | 6 | 11
  Sex, Unknown | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 10 | 3 | 13
  Not Hispanic or Latino | 11 | 3 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 6 | 1 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 9 | 13 | 27
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 18 | 42
Role [Count of Participants; unit: Participants]
  Pharmacist | 0 | 0 | 10 | 10
  Pharmacy technician | 4 | 0 | 5 | 9
  Pharmacy assistant | 0 | 0 | 2 | 2
  pharmacy director | 0 | 0 | 1 | 1
  pharmacist-in-charge | 3 | 0 | 0 | 3
  Staff pharmacist | 4 | 0 | 0 | 4
  Parents | 0 | 13 | 0 | 13
Years in practice (pharmacist only) [Mean (Standard Deviation); unit: years] — Population: This measure was only assessed for participants identifying as pharmacists.
  years
    number analyzed (Participants) | 7 | 0 | 18 | 25
    (all) | 7.4 (7) |  | 19.22 (17.13) | 13.31 (8.36)
Years working in pharmacy (other personnel) [Mean (Standard Deviation); unit: years] — Population: This measure of was only assessed for Aim 2 participants.
  years
    number analyzed (Participants) | 0 | 0 | 18 | 18
    (all) |  |  | 11.88 (6.83) | 11.88 (6.83)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Providing HPV Vaccination to Children and of the Proposed Communication Strategy to Support HPV Vaccination
Description: The survey was developed by study researchers based upon the Implementation Outcomes Questionnaire (IOQ) (Livet M, et al. 2021.). It was used to capture change of participants' perceptions pre/post training. There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point Likert scale indicate greater level of agreement that the intervention was acceptable to support HPV vaccination delivery to children ages 9-17. We calculated the average scale based on numeric scores. For questions that were asked in a reverse fashion, we reversed the score accordingly.
Time Frame: Up to 6 months after baseline survey and communication training
Population: This outcome measure was only assessed for Aim 2 participants. Only Aim 2 participants who completed all required Aim 2 protocol activities were assessed for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PROMOTE Intervention (Aim 2)
Number analyzed (Participants) | 13
units on a scale | 4.1 (0.664)

2. Primary Outcome: Appropriateness of Providing HPV Vaccination to Children and of the Proposed Communication Strategy to Support HPV Vaccination
Description: The survey was developed by study researchers based upon the Implementation Outcomes Questionnaire (IOQ) (Livet M, et al. 2021.). It was used to capture change of participants' perceptions pre/post training. There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point scale indicate greater level of agreement that the intervention was appropriate to support HPV vaccination delivery to children ages 9-17. We calculated the average scale based on numeric scores. For questions that were asked in a reverse fashion, we reversed the score accordingly.
Time Frame: Up to 6 months after baseline survey and communication training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PROMOTE Intervention (Aim 2)
Number analyzed (Participants) | 13
units on a scale | 4.0 (0.502)

3. Primary Outcome: Feasibility of Providing HPV Vaccination to Children and of the Proposed Communication Strategy to Support HPV Vaccination
Description: The survey was developed by study researchers based upon the Implementation Outcomes Questionnaire (IOQ) (Livet M, et al. 2021.). It was used to capture change of participants' perceptions pre/post training. There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point scale indicate greater level of agreement that the intervention was feasible to support HPV vaccination delivery to children ages 9-17. We calculated the average scale based on numeric scores. For questions that were asked in a reverse fashion, we reversed the score accordingly.
Time Frame: Up to 6 months after baseline survey and communication training
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PROMOTE Intervention Aim 2: Participants in the intervention group an adapted multi-modal communication strategy to support HPV vaccination in pharmacies administered by the Principal Investigator. Participants are pharmacy staff in Western Washington.
  The intervention consists of a multi-modal strategy that includes adapting an existing electronic "forecasting" system to identify vaccine eligible children who are due for vaccination and communication training for pharmacy staff to effectively recommend HPV vaccination.
  The intervention was delivered in one 60-minute session recorded and available online as a continuing education training that covered five modules: 1) educational overview of adolescent vaccination, 2) overview of the communication strategy, 3) process for integrating the strategy into clinical workflow, 4) training on communication strategy, and 5) pharmacy staff practice of the strategy.
Arm/Group | PROMOTE Intervention Aim 2
Number analyzed (Participants) | 13
units on a scale | 4.1 (0.529)

4. Primary Outcome: Self-efficacy of Providing HPV Vaccination
Description: The survey was developed by study researchers and included validated measures from a 31-item medication therapy management (MTM) efficacy scale (Martin B, et al. 2010) and a statewide survey of healthcare providers (McRee AL, et.al. 2014). It was used to capture change of participants' perceptions pre/post training. For this outcome there were five answers to each survey question reflecting how confident the respondent is in performing tasks related to providing HPV vaccinations to children, and each answer is given a score from 1 to 5, with 1 being not at all confident/strongly disagree and 5 being completely confident/strongly agree. Higher numerical scores on the 5-point scale reflect higher levels of self-efficacy or confidence in personal ability to complete vaccination process actions. We calculated the average scale based on numeric scores.
Time Frame: Baseline (pre-intervention) and up to 6 months following receipt of one 60-minute training session (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PROMOTE Intervention (Aim 2)
Number analyzed (Participants) | 13
units on a scale
  vaccine administration tasks (pre) | 4.2 (0.893)
  vaccine administration tasks (post) | 4.3 (0.798)
  personal interactions (pre) | 2.8 (0.830)
  personal interactions (post) | 3.4 (0.919)
  goal setting (pre) | 2.7 (0.983)
  goal setting (post) | 3.5 (1.107)
  HPV vaccine hesitancy (pre) | 2.6 (0.941)
  HPV vaccine hesitancy (post) | 3.3 (1.045)
Statistical Analysis 1: Comparison: PROMOTE Intervention (Aim 2); Test type: Other; 2-sided t-test conducted for pre- and post-training results

5. Primary Outcome: Adoption of HPV Vaccination
Description: Will conduct audits of the pharmacy electronic records to assess adoption of HPV vaccination, measured as the total sum (count) of HPV vaccinations administered by all eligible Aim 2 pharmacists.
Time Frame: Baseline (pre-intervention) and up to 6 months following receipt of one 60-minute training session (post-intervention)
Population: vaccine administration data for pharmacists who were participating in the study, pre and post-intervention. This outcome measure was only assessed for Aim 2 participants. Only Aim 2 participants who completed all required Aim 2 protocol activities were assessed for this measure.
Measure: Number; unit: sum of vaccine doses administered
Groups:
- PROMOTE Intervention: Participants in the intervention group an adapted multi-modal communication strategy to support HPV vaccination in pharmacies administered by the Principal Investigator. Participants are pharmacy staff in Western Washington.
  The intervention consists of a multi-modal strategy that includes adapting an existing electronic "forecasting" system to identify vaccine eligible children who are due for vaccination and communication training for pharmacy staff to effectively recommend HPV vaccination.
  The intervention was delivered in one 60-minute session recorded and available online as a continuing education training that covered five modules: 1) educational overview of adolescent vaccination, 2) overview of the communication strategy, 3) process for integrating the strategy into clinical workflow, 4) training on communication strategy, and 5) pharmacy staff practice of the strategy.
Arm/Group | PROMOTE Intervention
Number analyzed (Participants) | 13
sum of vaccine doses administered
  pre-intervention | 2
  post-intervention | 20
Statistical Analysis 1: Comparison: PROMOTE Intervention; Test type: Other; We grouped pharmacy data on vaccines delivered pre/post intervention into six categories: HPV vaccine, Tdap, Meningococcal, Influenza, COVID-19, and other vaccines. We then compared the counts of total vaccines that were conducted in each group pre- and post-training

6. Primary Outcome: Adoption of Other Adolescent Vaccines
Description: Will conduct audits of the pharmacy electronic records to assess adoption of other adolescent vaccination, measured as the total sum (count) of adolescent vaccinations administered by all eligible Aim 2 pharmacists.
Time Frame: Baseline (pre-intervention) and up to 6 months following receipt of one 60-minute training session (post-intervention)
Population: vaccines administered by pharmacists participating in the study, pre- and post-intervention. This outcome measure was only assessed for Aim 2 participants. Only Aim 2 participants who completed all required Aim 2 protocol activities were assessed for this measure.
Measure: Number; unit: sum of vaccine doses administered
Arm/Group | PROMOTE Intervention
Number analyzed (Participants) | 13
sum of vaccine doses administered
  pre-intervention | 75
  post-intervention | 145
Statistical Analysis 1: Comparison: PROMOTE Intervention; Test type: Other; [other analysis details as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected/assessed.
Description: Adverse events were not collected/assessed.
Arm/Group | PROMOTE Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04660331/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04660331/ICF_000.pdf